CLINICAL TRIAL: NCT03261609
Title: Risk of Chronic Diseases in Young Adults Born Preterm: Relationship With Inflammation and Oxidative Stress Biomarkers.
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Jewish General Hospital (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Anne Monique NUYT,MD, MD, Professor of Pediatrics, St. Justine's Hospital
Other Study IDs: HAPI clinical project
Record Dates: First submitted 2017-07-28; First posted 2017-08-25 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Prematurity; Extreme
Keywords: extremely preterm; young adults; CVD risks factors; inflammation; chronic health conditions; term
MeSH Terms: conditions — Premature Birth; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The team collected the blood and urine of the participants. They kept whole blood and urine the the biobank. The group also isolated the plasma and serum to perform assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extremely preterm (EPT): All adults born at gestational age (GA) <29 wks at CHU Sainte-Justine (CHUSJ), the Royal Victoria Hospital (RVH), and the Jewish General Hospital (JGH), Montreal, in 1987-97.
  Inclusion criteria: (a) Birth at GA<29 wks, (b) age 18-29 years at the time of assessment (age of peak human physiological function).
  Exclusion criteria: (a) currently pregnant due to X-ray related risks, (b) severe neurosensory deficit preventing test completion. In case of twins (or +), if both fulfil inclusion criteria, only one will selected (random) to participate to the study.
  Interventions: Other: preterm birth
- Term or controls: Same-sex friends identified by EPT subject who have accepted to be contacted. Inclusion criteria: (a) Birth at GA ≥37 wks, (b) born in Quebec, to account for health care access during pregnancy and throughout infancy/childhood, (c) birth date within 2 years of index case, (d) age 18-29 years at the time of assessment, (e) same self-reported race as preterm participant.
  Exclusion criteria: (a) currently pregnant due to X-ray related risks, (b) severe neurosensory deficit preventing test completion.
  Interventions: Other: preterm birth

INTERVENTIONS:
Other: preterm birth — The study compares young adult subjects born premature (< 29 weeks) versus term (-> 37 weeks)

SUMMARY:
The purpose of the HAPI project is to study the overall health of preterm infants once they reach adulthood. The investigators would like to compare the health of adults born preterm with that of adults born full-term. They would also like to find the early signs, or biomarkers, of chronic diseases such as high blood pressure, diabetes, osteoporosis, and chronic lung diseases.

Such biomarkers would allow for early diagnosis and prevention. Furthermore, the investigators would like to understand why some people born preterm are more likely to develop chronic disease. They believe that inflammation and oxidative stress may play a part. Oxidative stress is present when the body is not able to defend itself against oxygen-derived products that can damage our cells.

To carry out this study, the investigators will examine 6 aspects of the health: (1) heart and circulation, (2) kidneys, (3) lungs, (4) metabolism - sugars and fats in the blood, (5) bones, and (6) eyes.

DETAILED DESCRIPTION:
The participants, from both groups will spend a whole day at St. Justine's hospital. Upon arrival after an overnight fast, vital signs and anthropometric measures are taken. Then blood and urine are obtained as well and a pregnancy test is performed for women. After inserting a intravenous catheter, around 55 mL of blood is taken and sent to the biochemistry department and to our laboratory. A oral glucose tolerance test is also performed with blood sampling over 2hours.

Then a renal and carotid ultrasounds, as well as a osteodensitometry test (bone mineral density and body muscle/fat composition) are done. Ophtalmology exam is realized by ophtalmologist, including visual acuity, contrast and fundus photograph, then the participants are provided with a standardized light lunch.

A thorough cardiac ultrasound, as well as assessment of major arteries (aorta, carotid, brachial) structure and function are performed. Pulmonary function tests are done before a fitness test for VO2 max, and repeated with bronchodilatator after the fitness test.

Prior to leaving, participants are given a ambulatory blood pressure monitor for them to carry for 24 consecutive hours over the following 2 days.

Prior to the study day, participants are sent questionnaires to be filled in advance by themselves and by each of their parent. During the study day, other questionnaires regarding their lifestyles and medical condition are also filled. Overall, information is obtained about:

(1) Socio-economic status: Occupation, education level and income of participant and parents. (2) Family history: Parental health (including maternal pregnancies) and familial (1st and 2nd degree) premature history of cardiovascular diseases (CVD), type-2 diabetes, chronic pulmonary or renal diseases. (3) Personal medical history: Current medication use (including anti-inflammatory medications), medical history, current symptoms, and growth parameters from birth to present (according to medical records and child health care booklet), age at menarche.

(4) Health-related behaviors: (a) regular physical activities (Minnesota and Huet validated questionnaires) (b) Smoking and alcohol consumption. (c) Diet assessed through the validated and self-administered 73-item Food Frequency Questionnaire (FFQ). (d) SF-36 Health Survey.

In addition to the study protocol, the subjects are invited to contribute extra biosamples to our blood (3 ml) and urine (1 ml) biobank.

ELIGIBILITY:
Inclusion Criteria:

EPT :

* Birth at GA<29 wks
* Age 18-29 years at the time of assessment (age of peak human physiological function)

Terms:

* Birth at GA ≥37 wks
* Born in Quebec, to account for health care access during pregnancy and throughout infancy/childhood
* Birth date within 2 years of index case
* Age 18-29 years at the time of assessment
* Same self-reported race as preterm participant.

Exclusion Criteria:

Both groups :

* Currently pregnant due to X-ray related risks
* Severe neurosensory deficit preventing test completion.
* In case of twins (or +), if both fulfil inclusion criteria, only one will selected (random) to participate to the study

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The extremely preterm subjects need to come with a same sex born term subject.
Study Population: All adults born at GA<29 wks at CHU Sainte-Justine, the Royal Victoria Hospital, and the Jewish General Hospital, Montreal, in 1987-97. For each EPT subject, a friend control matched on sex is selected to control in part for lifestyle and social factors (e.g. diet, physical activity, health care visits), and environmental exposure that may affect inflammatory status and disease risk. Indeed, given the known link between lower socio-economic status, lifestyle habits and CVD risk factors, and that women from lower SES and with poor lifestyle behaviors are at increased risk to deliver prematurely, a friend control, who is more likely to have evolved in a similar milieu, will allow us to better isolate the effect of preterm birth on studied outcomes from socio-environmental factors.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-04-29 (Actual)

PRIMARY OUTCOMES:
Markers of inflammation | 1 hour
  Blood samples for measurements of biomarkers of inflammation are collected in the morning the day of the visit. Monocyte chemoattractant-1 (pg/mL), Interleukine-6 (pg/mL), tumor necrosis factor-alpha (pg/mL), intercellular adhesion molecule-1 (pg/mL), vascular cell adhesion molecule-1 (pg/mL), high-sensitivity C-reactive protein (pg/mL).
Markers of oxydative stress in the blood | 1 hour
  Blood samples for measurements of biomarkers of oxidative stress are collected in the morning the day of the visit. Blood : Glutathione (GSH and GSSG (nmol/mg of proteins)) and Redox potential using the Nernst equation and the values of GSH and GSSG (mV).
Markers of oxydative stress in the urine | 1 hour
  Urine 8-prostaglandin F2-alpha (pg/mL).
Markers of oxydative stress in the plasma | 1 hour
  Oxidized LDL (U/L)

SECONDARY OUTCOMES:
CVD risk factors and indicators of (sub)clinical disease: blood pressure | 1 hour
  Blood pressure (mmHg)
CVD risk factors and indicators of (sub)clinical disease: Cardiac structure and function by echocardiography- LV hypertrophy #1 | 30 min
  Cardiac structure and function by echocardiography. Left ventricle hypertrophy determined by the LV mass (g) indexed to body surface area (BSA in m2) giving a unit of g/m2.
CVD risk factors and indicators of (sub)clinical disease: Cardiac structure and function by echocardiography- LV hypertrophy #2 | 30 min
  Cardiac structure and function by echocardiography. Left ventricle hypertrophy determined by the interventricular septum thickness (cm).
CVD risk factors and indicators of (sub)clinical disease: Cardiac structure and function by echocardiography -LV hypertrophy #3 | 30 min
  Cardiac structure and function by echocardiography. Left ventricle hypertrophy determined by LV dysfunction (%) or by endocardial fractional shortening (%)
CVD risk factors and indicators of (sub)clinical disease: Arterial structure and function by ultrasound. | 1 hour
  Arterial structure and function (mm) will be measured using a Dopller ultrasound.
CVD risk factors and indicators of (sub)clinical disease: Adiposity measures #1 | 15 min
  Body mass index in kg/m2, calculating using the weight in kg and the height in m
CVD risk factors and indicators of (sub)clinical disease: Adiposity measures #2 | 30 min
  Using lean and fat body (g) m
CVD risk factors and indicators of (sub)clinical disease: glucose homeostasis | 2 hours
  Plasma fasting glucose (mmol/L) and insulin (mmol/L) and different times after a 75 g of glucose load.
CVD risk factors and indicators of (sub)clinical disease: Fasting lipid profile | 1 hour
  Plasma triglycerides (mmol/L), HDL (mmol/L) and LDL (mmol/L).
CVD risk factors and indicators of (sub)clinical disease: kidneys functions #1 | 30 min
  Urinary protein excretion (albumin/creatinine ratio, mg/mmol), eGFR cystatin C (cystatin C : mg/L) (mL/min/1.73 m2). The formula use the cystatin C values in mg/mL, the standardized serum cystatin min and max, the age (in years) and the sex (female: 0.932, male : 1).
CVD risk factors and indicators of (sub)clinical disease: kidneys functions #2 | 15 min
  Use of the eGFR cystatin C formula (cystatin C : mg/L) (mL/min/1.73 m2). The formula use the cystatin C values in mg/mL, the standardized serum cystatin min and max, the age (in years) and the sex (female: 0.932, male : 1).
CVD risk factors and indicators of (sub)clinical disease: pulmonary functions #1 | 30 min
  FEV (%)
CVD risk factors and indicators of (sub)clinical disease: pulmonary functions #2 | 30 min
  Airflow obstruction (FEV1/FVC ratio, no units).
CVD risk factors and indicators of (sub)clinical disease: Questionnaires #1 | 2 hours
  Determinants of health. Questionnaires about socio-economics status, family history, personal medical history.
CVD risk factors and indicators of (sub)clinical disease: Questionnaires #2 | 2 hours
  Determinants of health. Maternal obstetrical and subjects neonatal history.
CVD risk factors and indicators of (sub)clinical disease: Questionnaires #3 | 2 hours
  Determinants of health. Health-related behaviors
CVD risk factors and indicators of (sub)clinical disease: Questionnaires #4 | 2 hours
  Determinants of health. Food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anne Monique Nuyt, MD, Principal Investigator — St. Justine's Hospital; Thuy Mai Luu, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- StJustine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: Starting 1 year after all results of the study are published.
Access Criteria: Request of collaboration through data access will be examined by the PI's.

REFERENCES:
- [Derived] Ravizzoni Dartora D, Flahault A, Pontes CNR, He Y, Deprez A, Cloutier A, Cagnone G, Gaub P, Altit G, Bigras JL, Joyal JS, Mai Luu T, Burelle Y, Nuyt AM. Cardiac Left Ventricle Mitochondrial Dysfunction After Neonatal Exposure to Hyperoxia: Relevance for Cardiomyopathy After Preterm Birth. Hypertension. 2022 Mar;79(3):575-587. doi: 10.1161/HYPERTENSIONAHA.121.17979. Epub 2021 Dec 28. PMID 34961326
- [Derived] Dartora DR, Flahault A, Luu TM, Cloutier A, Simoneau J, White M, Lapointe A, Villeneuve A, Bigras JL, Altit G, Nuyt AM. Association of Bronchopulmonary Dysplasia and Right Ventricular Systolic Function in Young Adults Born Preterm. Chest. 2021 Jul;160(1):287-296. doi: 10.1016/j.chest.2021.01.079. Epub 2021 Feb 5. PMID 33549599
- [Derived] Gervais AS, Flahault A, Chan T, Bastien-Tardif C, Al-Simaani A, Cloutier A, Luu TM, Abadir S, Nuyt AM. Electrocardiographic features at rest and during exercise in young adults born preterm below 30 weeks of gestation. Pediatr Res. 2020 Aug;88(2):305-311. doi: 10.1038/s41390-020-0814-9. Epub 2020 Mar 2. PMID 32120379
- [Derived] Flahault A, Paquette K, Fernandes RO, Delfrate J, Cloutier A, Henderson M, Lavoie JC, Masse B, Nuyt AM, Luu TM; HAPI collaborating group*. Increased Incidence but Lack of Association Between Cardiovascular Risk Factors in Adults Born Preterm. Hypertension. 2020 Mar;75(3):796-805. doi: 10.1161/HYPERTENSIONAHA.119.14335. Epub 2020 Jan 27. PMID 31983307
- [Derived] Paquette K, Fernandes RO, Xie LF, Cloutier A, Fallaha C, Girard-Bock C, Mian MOR, Lukaszewski MA, Masse B, El-Jalbout R, Lapeyraque AL, Santos RA, Luu TM, Nuyt AM. Kidney Size, Renal Function, Ang (Angiotensin) Peptides, and Blood Pressure in Young Adults Born Preterm. Hypertension. 2018 Oct;72(4):918-928. doi: 10.1161/HYPERTENSIONAHA.118.11397. PMID 30354721